CLINICAL TRIAL: NCT01011088
Title: Paternal Psychosis Evaluation After First Baby Born
Brief Title: Paternal Psychosis After Baby Born
Acronym: PAPABAB
Status: Completed | Type: Observational
Sponsor: Nanjing Medical University (Other)
Responsible Party: XiaoFeng Shen, Nanjing Medical University
Other Study IDs: NMU-200911-MZ018; NJFY09331M012 (Other Grant/Funding Number: Nanjing Medical University)
Record Dates: First submitted 2009-11-09; First posted 2009-11-11 (Estimated); Last update posted 2010-06-04 (Estimated); Status verified 2010-06

CONDITIONS: Psychosis
Keywords: Paternity; Psychology; Risk factor
MeSH Terms: conditions — Psychotic Disorders

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Early phase: Psychoses within the first 3 months after baby born
- Delayed phase: Psychoses > 3 months to one year after baby born

INTERVENTIONS:
Other:  — Not any artificial interventions were given

SUMMARY:
A large number of studies have investigated the psychological disorders occurred in postpartum women, and found that postpartum psychosis is common in new mothers.

However, the situation of paternal psychological status after they had their first baby is not assessed. The investigators hypothesized that they had a high occurrence of paternal psychosis after first baby born. In addition, different factors might influence its onset and development in new fathers.

ELIGIBILITY:
Inclusion Criteria:

* Men will be the would-be fathers
* Chinese

Exclusion Criteria:

* Age < 18 years or > 50years
* Not willing to participating or completing the whole study at any time

Ages: 19 Years to 49 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Study Population: Fathers with their first baby born
Sampling Method: Probability Sample
Enrollment: 387 (Actual)
Dates: Start 2009-11; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Incidence of psychoses | Within the first 90 days and 90 days to 12 months postpartum

SECONDARY OUTCOMES:
Economic level before baby born | One year before baby born
Social status before baby born | One year before baby born
Psychological level before baby born | From birth of the fathers to the time of their baby born,this is varing from different fathers and received by history records
Maternal intrapartum complications | From the onset of painful labor (0 min of delivery) to the completion of birth (varying in different women and/or different labor procedures)
Baby characteristics | One minute, 5min, 15min after baby was born

CONTACTS AND LOCATIONS:
Overall Officials: XiaoFeng Shen, MD, Study Director — Nanjing Medical University
Locations (1):
- Nanjing Maternity and Child Health Care Hospital, Nanjing, Jiangsu, China